CLINICAL TRIAL: NCT00388076
Title: A Phase I, Open-Label, Study of the Safety, Tolerability, and Pharmacokinetics of Pazopanib in Combination With Paclitaxel on a Weekly Schedule for Three Consecutive Weeks of a 28-Day Cycle, Paclitaxel and Carboplatin on an Every 21 Days Schedule and Lapatinib and Paclitaxel on a Weekly Schedule for Three Consecutive Weeks of a 28- Day Cycle
Brief Title: Pazopanib (VOTRIENT) Plus Paclitaxel (TAXOL), Pazopanib Plus Paclitaxel (TAXOL) Plus Carboplatin (PARAPLATIN), and Pazopanib Plus Paclitaxel (TAXOL) Plus Lapatinib (TYKERB)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG105427
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: carboplatin; lapatinib; TAXOL; PARAPLATIN; paclitaxel; TYKERB; Pazopanib
MeSH Terms: conditions — Breast Neoplasms | interventions — pazopanib; Lapatinib; Paclitaxel; Carboplatin

ARMS (3):
- Part 1 (Experimental): pazopanib and paclitaxel
  Interventions: Drug: Pazopanib; Drug: paclitaxel
- Part 2 (Experimental): pazopanib, paclitaxel, and carboplatin
  Interventions: Drug: Pazopanib; Drug: paclitaxel; Drug: carboplatin
- Part 3 (Experimental): pazopanib, paclitaxel, and lapatinib
  Interventions: Drug: Pazopanib; Drug: Lapatinib; Drug: paclitaxel

INTERVENTIONS:
Drug: Pazopanib — pazopanib in combination with paclitaxel in Part 1, paclitaxel and carboplatin in Part 2, and paclitaxel and lapatinib in Part 3
Drug: Lapatinib — Lapatinib in combination with pazopanib and paclitaxel in Part 3
  Arms: Part 3
Drug: paclitaxel — in combination with pazopanib
  Other Names: TAXOL
Drug: carboplatin — in combination with pazopanib
  Other Names: PARAPLATIN
  Arms: Part 2

SUMMARY:
Pazopanib will be given with TAXOL in one part, in another part pazopanib will be given with TAXOL and PARAPLATIN, and in a third part pazopanib will be given with TAXOL and lapatinib (patients separated in each part). Toxicity monitoring will enable us to find the largest dose of pazopanib daily that can be safely given in combination with the chemotherapy agents TAXOL and PARAPLATIN, and with lapatinib, as well as what side effects are likely to manifest when these agents are given together and whether the combination of pazopanib with chemotherapy, helps to treat different types of cancer. Another objective is to find out how much pazopanib, TAXOL, PARAPLATIN and lapatinib are in the blood at specific times after the agents are given. Collecting the blood samples requires that the patients remain in the vicinity of the clinic overnight on 2 occasions.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of cancer, except cervical cancer
* Eastern Cooperative Oncology Group performance Status of 0 or 1
* Peripheral neuropathy of Grade 1 or less
* Adequate bone marrow function (absolute neutrophils, platelets and hemoglobin levels as per protocol)
* Adequate renal function as per protocol
* Urine creatinine ratio as per protocol
* Adequate hepatic function as per protocol
* Coagulation tests as per protocol
* Male of female at least 18 years of age
* A woman is eligible to enter and participate in the study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any woman who:
* Has had a hysterectomy,
* Has had a bilateral oophorectomy (ovariectomy),
* Has had a bilateral tubal ligation,
* Is post-menopausal (total cessation of menses for at least 1 year)
* Childbearing potential, has a negative serum or urine pregnancy test at screening, and agrees to one of the following:
* An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the patient's entry and is the sole sexual partner for that woman.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, throughout the clinical trial, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR male condom and diaphragm.
* Predicted life expectancy of at least 12 weeks
* Written informed consent
* Able to swallow and retain oral medications.

Exclusion criteria:

* No more than 3 prior lines of cytotoxic chemotherapy for metastatic disease are allowed.
* No major surgery, nor cytotoxic chemotherapy, investigational agents, or radiotherapy within the last 28 days and subject must have recovered fully from whatever their last treatment was at the time of enrollment.
* Women who are pregnant or breast feeding are not eligible to enroll.
* Cannot have poorly controlled hypertension.
* Cannot have corrected QT (QTc) prolongation
* Cannot have Class III or IV heart failure as defined by the New York Heart Association functional classification system.
* Cannot have arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within the last 3 months.
* Cannot use of therapeutic warfarin.
* Cannot have history of bleeding (hemoptysis, hematuria, GI blood loss, epistaxis, or others with greater than Grade 1 according to CTC Criteria) within six weeks prior to beginning therapy or any clinical indications of current active bleeding or bleeding diathesis.
* Cannot have history or clinical evidence of CNS metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 2 months prior to beginning study treatment.
* Cannot have any serious and/or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with patient safety or obtaining consent.
* Cannot have history of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism or excretion of pazopanib, paclitaxel, or carboplatin. Has any unresolved bowel obstruction or diarrhea. Has clinically significant gastrointestinal abnormalities that may increase the risk for GI bleeding including, but not limited to:

  * active peptic ulcer disease,
  * known intraluminal metastatic lesion(s) with suspected bleeding,
  * inflammatory bowel disease including ulcerative colitis, or other GI conditions with increased risk of perforation,
  * history of abdominal fistula, GI perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Subject must not have psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Subject must not take any specifically prohibited medication specified in the protocol during the study or requires any of these medications during treatment with pazopanib.
* Subject must not have clinical history, current alcohol or illicit drug use which, in the judgment of the Investigator, would interfere with the patient's ability to comply with the dosing schedule and protocol-specified evaluations.
* Subject must not be allergic to either TAXOL or PARAPLATIN, or any other taxane or platinum containing compound.
* Subject must not have a current diagnosis of cervical cancer.
* Subject must not have known endobronchial metastasis or involvement of large pulmonary vessel(s) by tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-04-28 (Actual); Primary Completion 2009-07-21 (Actual); Study Completion 2009-07-21 (Actual)

PRIMARY OUTCOMES:
Adverse Effects, Laboratory parameters | before and after taking the study medications.

SECONDARY OUTCOMES:
Blood samples | over a 24 hour period
Tumors | will be measured at routine intervals throughout (e.g. by CT scan).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Nashville, Tennessee

REFERENCES:
- [Background] Burris HA 3rd, Dowlati A, Moss RA, Infante JR, Jones SF, Spigel DR, Levinson KT, Lindquist D, Gainer SD, Dar MM, Suttle AB, Ball HA, Tan AR. Phase I study of pazopanib in combination with paclitaxel and carboplatin given every 21 days in patients with advanced solid tumors. Mol Cancer Ther. 2012 Aug;11(8):1820-8. doi: 10.1158/1535-7163.MCT-11-0997. Epub 2012 Jun 7. PMID 22679111
- [Background] Tan AR, Dowlati A, Jones SF, Infante JR, Nishioka J, Fang L, Hodge JP, Gainer SD, Arumugham T, Suttle AB, Dar MM, Lager JJ, Burris HA 3rd. Phase I study of pazopanib in combination with weekly paclitaxel in patients with advanced solid tumors. Oncologist. 2010;15(12):1253-61. doi: 10.1634/theoncologist.2010-0095. Epub 2010 Dec 8. PMID 21147873
- [Derived] Tan AR, Dowlati A, Stein MN, Jones SF, Infante JR, Bendell J, Kane MP, Levinson KT, Suttle AB, Burris HA 3rd. Phase I study of weekly paclitaxel in combination with pazopanib and lapatinib in advanced solid malignancies. Br J Cancer. 2014 May 27;110(11):2647-54. doi: 10.1038/bjc.2014.233. Epub 2014 May 6. PMID 24800949
- See also: Results for study VEG105427 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG105427?search=study&study_ids=VEG105427#rs